CLINICAL TRIAL: NCT03846024
Title: Orthosis of Acute Traumatic Rib Fractures Via RibFx Belt for Pain Alleviation and Improved Pulmonary Function: A Pre-Post Interventional Trial for Quality Improvement
Brief Title: Orthosis of Acute Traumatic Rib Fractures Via RibFx Belt for Pain Alleviation and Improved Pulmonary Function
Acronym: RibFx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impact of COVID-19 pandemic on COVID precautions and restrictions of research in the clinical setting; challenges with participant engagement and data collection post-discharge.
Sponsor: University of Vermont Medical Center (Other)
Collaborators: PelvicBinder, Inc. (Industry)
Responsible Party: Principal Investigator, Ajai K Malhotra, MD FACS, Chief, Acute Care Surgery Division, University of Vermont Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB CHRMS 18-0646
Record Dates: First submitted 2018-12-15; First posted 2019-02-19 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Rib Fracture; Rib Fracture Multiple; Trauma; Trauma Chest; Trauma Injury; Trauma, Multiple
Keywords: RibFx; PelvicBinder; Rib Fractures; Trauma; Pulmonary toilet; Incentive Spirometry
MeSH Terms: conditions — Rib Fractures; Wounds and Injuries; Thoracic Injuries; Accidental Injuries; Multiple Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RibFx belt arm (Experimental): Each patient in the interventional arm will be fitted with a RibFx orthosis belt, which is to be worn during the majority of their day (excluding showering/bathing). It will be encouraged (though not mandatory) to wear at night. Patients in both the control and interventional arm will be expected to participate in pulmonary hygiene / toilet exercises with guided and independent incentive spirometry as per our normal routine and standard of care. There are no other interventions or procedures that the patients will be subjected to for the research trial- other procedures/interventions will be performed only if the clinical care team feels they are indicated.
  Interventions: Device: RibFx Orthosis Belt
- Control (No Intervention): Patients in the control arm receive normal standard of care for rib fractures at the participating institution.
  The current standard of care for rib fractures at the University of Vermont (participating institution) is as follows: includes oral and IV analgesia and other multimodal pain control as appropriate, including muscle relaxants such as methocarbamol (robaxin) unless there is a contraindication, pulmonary hygiene/toilet and respiratory care (including frequent evaluations by physicians, respiratory therapists, and nursing staff, early mobilization, and monitoring for pulmonary complication (via vital signs, pulse oximetry, oxygen requirement, chest imaging if appropriate).

INTERVENTIONS:
Device: RibFx Orthosis Belt — Each patient in the interventional arm will be fitted with a RibFx orthosis belt, which is to be worn during the majority of their day (excluding showering/bathing). It will be encouraged (though not mandatory) to wear at night. Patients in both the control and interventional arm will be expected to participate in pulmonary hygiene / toilet exercises with guided and independent incentive spirometry as per our normal routine and standard of care. There are no other interventions or procedures that the patients will be subjected to for the research trial- other procedures/interventions will be performed only if the clinical care team feels they are indicated.
  Arms: RibFx belt arm

SUMMARY:
Acute traumatic rib fractures are a common issue for patients of trauma surgeons. They inflict substantial morbidity, the most dreaded and consequential of which are pulmonary complications. While these fractures are often treated non-operatively, there is a continued need for effective adjuvant treatments to improve rib fracture pain and outcomes. Prior studies have evaluated outcome measures for traumatic rib fractures that include respiratory failure, tracheostomy requirement, ICU length of stay, hospital length of stay, narcotic requirement, daily maximum incentive spirometry volume, pneumonia, and mortality .

Rib belts, which have been present since at least 1945, have long been used to provide pain relief via chest wall stabilization [3]. However there is an extreme paucity of literature regarding their clinical efficacy, and their use has largely been abandoned due to concerns that they may have been overly constricting and resulted in poorer respiratory (pulmonary/breathing) outcomes. Newer generation rib belts are more elastic and theoretically less constricting than their earlier generation predecessors, however their clinical efficacy has not been yet demonstrated. The investigators will therefore plan to perform a prospective trial to determine if these rib strapping devices are effective clinical tools in the traumatic rib fracture population. The goal of the study is institutional quality improvement, to determine if the investigators see benefit of these devices for the pain management of our trauma population. The investigators will also conduct this as a pilot trial for hopeful future research applications, however the overall goal is institutional improvement.

Patients determined to be eligible for the study by the admitting physician (and per the previously defined criteria) will be recruited to enroll in the project within the first 24 hours of their hospital admission. Recruited patients will be offered the opportunity to consent to enrollment in the study and will be assigned by the study team into either the intervention (RibFx belt +current standard of care) or control (current standard of care) arm in a quasi-experimental prospective design: untreated control group with dependent pretest and posttest samples. In this manner, the intervention arm will be both compared to themselves (pretest vs. posttests) as well as to a control group not exposed to the intervention.

The relevant study materials will be included in their paper (physical) and electronic chart. Patients upon enrollment in the study will undergo an initial assessment that will include their baseline pain scores, narcotic consumption, incentive spirometry scores, and the subjective self-reported results of their questionnaire (the pre-test questionnaire- see attached). Patients will continue to be scored on objective (incentive spirometry results, opioid pain medicine consumption) and subjective variables (pain scores) during their hospital course. Between 24-48 hours after enrollment, they will be prompted to again complete a similar 2nd questionnaire post-test (if they are discharged from the hospital at this point in the time course, they will be sent home with the questionnaire and prompted to complete it at home). At their follow up appointment in trauma clinic (which will be coordinated by the research team to be as close as possible to 3 weeks post injury), they will have the opportunity to again voluntarily complete a final short questionnaires (post-test) that assess their pain control and respiratory function over the last 3 weeks. At this point, their involvement in the trial will be complete.

Patients themselves will play an active role in data collection during the trial, and will be instructed and prompted in how to do so. Patients will be expected to fill out a worksheet on a daily basis, both while inpatient and after discharge, on their daily incentive spirometry scores as well as their minimum and maximum pain scale scores. This will be used to supplement the survey or questionnaire data, as well as the objective data from the electronic medical record.

The investigators will ultimately compare groups using a quasi-experimental design as follows: Untreated control group with dependent pretest and posttest samples. This will allow for a direct comparison of patient to patient within the intervention arm (patient pretest result serving as control compared to posttest result) . To observe for temporal variability, their will be a control group with no intervention as well (no rib belt worn) , however the principle aim of the study is the comparison of patients to themselves in a pre-test, post-test fashion.

DETAILED DESCRIPTION:
The purpose of this study is to ascertain whether the use of next generation rib orthosis belts (such as the RibFx) can improve patient outcomes following traumatic rib fractures within our population, whether it be by improving pain control, decreased respiratory complications, or increased patient satisfaction. The investigators hypothesize that the use of elastic rib belts will improve rib fracture pain control without compromising pulmonary function (statistically significant improvement in pain control without significant impairment in respiratory function or increase in respiratory complication). The investigators feel as though answering this question can help us as providers to improve the quality of care to our patients in our department.

Rib fractures are a common traumatic injury, and can cause substantial morbidity and mortality in the trauma population. As rib fractures most often are not treated with surgical intervention, there is demand for non-operative strategies to promote healing, pain control, and mechanical/musculoskeletal support. This can also help decrease the administration of potentially harmful pain medications such as opioid or narcotic pain medication. Further, as rib fracture pain can often be long lasting, this can truly increase quality of life for patients as they recover from these injuries.

The objectives of the clinical trial are to determine if rib orthosis via the use of the RibFx belt can improve patients after traumatic rib fractures by improving pain control without compromise of respiratory function or increase respiratory complications of rib fracture.

Per Jeffords Institute for Quality Data of the University of Vermont, there were 190 patients admitted the to Acute Care Surgery (Trauma) service at the University of Vermont Medical Center during the year 2016. Assuming that these numbers remain fairly static overtime as they have in the past, the investigators would expect approximately 16 patient admissions per month with the diagnosis of rib fracture (seasonal fluctuations do exist with more traumatic admissions during the summer months). The goal time period for the trial would be to conduct this trial during the summer, with a goal of 50 total patients. The investigators would therefore expect an enrollment period (data collection phase) of approximately 3 months.

During the study, appropriate patients will be recruited both to the control arm of the study and the intervention/comparison arm in a specified / non-randomized sequence as seen in the schematic below (First 5 patients control, next five patients intervention, next five patients control, next five patients intervention, next five patients control, final 25 patients intervention). Control arm will include 15 total patients. All will be consented to the study upon admission (first 24 hours of index hospitalization for injury) with full knowledge that they will either be undergoing no intervention other than receiving the current standard of care for rib fracture care per our institution's standard, and if assigned to the rib belt group, expected to wear the rib belt during their recovery.

The current standard of care for rib fractures at our institution is as follows: includes oral and IV analgesia and other multimodal pain control as appropriate, including muscle relaxants such as methocarbamol (robaxin) unless there is a contraindication, pulmonary hygiene/toilet and respiratory care (including frequent evaluations by physicians, respiratory therapists, and nursing staff, early mobilization, and monitoring for pulmonary complication (via vital signs, pulse oximetry, oxygen requirement, chest imaging if appropriate).

All patients will undergo initial "Pre-test" testing which will include baseline pain scores (1-10 traditional pain scale assessed every 8 hours, then averaged over the 24 hour period), initial narcotic consumption (in MME) for first 24 hours of hospitalization, maximum incentive spirometry score for first 24 hours of hospitalization, and pre-test questionnaire result (see attached questionnaire #1). As the study continues their relevant data will be collected, including both objective (incentive spirometry scores, opioid pain medication consumption, incidence of atelectasis and pneumonia) and subjective (pain scores, survey result) clinical data. Concurrently, The investigators will complete the trial with the intervention (RibFx belt) phase in which participants will be enrolled in the interventional arm of the study. The objective and subjective data will be collected in an identical fashion- the only difference between groups will be that this group will have been fitted with the RibFx belt for their hospital course and discharge.

The participants (both in the control and interventional groups) will again be asked to complete essentially the same brief surveys in a post-test fashion at two set time points: between 24-48 hours after initial enrollment in the study (Questionnaire #2)(if patient has been discharged at this point, they will be sent home with this survey and instructed when to complete), and at 3 weeks post-injury (this will be done at their clinic visit, assuming they are not still admitted to the hospital at this time point).

Patients will also be sent home with a work-book to record their incentive spirometry scores and pain scores (all patients will be sent home with an incentive spirometer, and all patients in the interventional group will be sent home with their Ribfx belt).

The following additional data will also be quantified from the medical record via manual data extraction: ICU length of stay, hospital length of stay, pulse oximetry and respiratory rate scores (taken from already collected vital signs every four hours), body mass index (BMI), bronchodilator (such as albuterol or other inhaled beta agonist) use, age, sex/gender, tobacco history/pack years, days on mechanical ventilator, narcotic requirement (in mean morphine equivalents or morphine equianalgesic dose per day).

In addition, an independent radiology physician will analyze the chest x-rays, CT chests of the patients enrolled in the study and grade them in a blinded fashion) on a scale for the following characteristics: Degree and quantity of rib fracture, presence and degree of atelectasis, presence of COPD/emphysematous change or other parenchymal lung disease, presence and degree of pneumothorax, bilateral vs. unilateral disease, presence of intrapleural fluid, evidence of "flail chest" segment, and presence of pulmonary contusion and other noted pathology (see the attached Radiology Grading Form document). The investigators will measure the degree of radiological severity and compare the control and interventional group to determine what differences in initial disease severity exist (so they can be accounted for).

Each patient in the interventional arm will be fitted with a RibFx orthosis belt, which is to be worn during the majority of their day (excluding showering/bathing). It will be encouraged (though not mandatory) to wear at night. Patients in both the control and interventional arm will be expected to participate in pulmonary hygiene / toilet exercises with guided and independent incentive spirometry as per our normal routine and standard of care. There are no other interventions or procedures that the patients will be subjected to for the research trial- other procedures/interventions will be performed only if the clinical care team feels they are indicated.

Patients will be assessed with three short questionnaires in a pretest , posttest fashion at both the onset of the study, 24-48 hours after enrollment, and at their follow-up appointment 3 weeks after (2 post test questionnaires). The initial evaluation will occur on initial assessment prior to placement of the rib belt (or, for the control/ non-intervention group, at the onset/first 24 hours of the study).

Each of the questionnaires is essentially the same with only brief modifications made in the first two questions to make them appropriate for the timing during the clinical course. However these are all attached (see Questionnaire 1,2,and 3).

Patients in both the intervention and control arms will present in post-admission follow up at a time period of 3 weeks post injury (range, 2-4 weeks) following their hospital admission, and will be asked to fill out a brief survey regarding their respiratory function and pain control. This survey will also inquire into compliance with the use of incentive spirometer, and compliance with the use of the RibFx belt (for patients in the intervention arm).

The surveys are a novel series of questionnaires using previously validated tools such as the COPD Assessment Test or CAT (Jones PW, Harding G, Berry P et al 2009) and the Brief Pain Inventory (BPI) in order to subjectively assess each patient's own breathing/ respiratory and pain symptoms. The surveys also have additional questions gaging their pain medication usage, compliance with their treatment therapies (including IS and rib belt usage, when applicable). The survey is designed to be completed in ten minutes. The survey was constructed with the assistance of a professor psychologist who specializes survey construction (Author ACB). There will be no financial compensation for survey completions.

All surveys will be adapted to apply to the unique population being surveyed- the post-trauma population. This may involve removal of some questions that are not applicable to the rib fracture patients. There are several questions on the questionnaire that might not be applicable to the control group- they are simply instructed to not complete those four questions.

The surveys have been modified in order to be more easily comprehended to the average patient, and to require minimal additional instruction (so that the patient can complete them independently with no additional prompting).

In this study, The investigators will utilize a quasi-experimental design to compare 35 subjects to themselves in a pre-test, post-test fashion. In addition, the investigators will have an additional 15 non-interventional control patients to observe for temporal changes in patient's symptoms not secondary to the intervention itself. However, it is important to note that the study is not powered to detect differences between the control group and the intervention group. The purpose of the control group is to observe for differences that occur in this population over time regardless of intervention (it should be assumed that pain will improve as time increases from the set injury point, regardless of intervention). Further, this preliminary data could potentially be used to calculate an accurate power calculation for a definitive randomized controlled trial.

Groups will be compared by demographical and clinical data to determine what potentially confounding differences exist between the arms of the study. Relevant objective data that will be used to determine group differences include (but not limited to): age, sex, tobacco use status (active/former/none), presence of asthma, presence of COPD, or presence of restrictive lung disease, home oxygen use, obstructive sleep apnea/ CPAP use, chronic pain incidence, narcotic/opioid medication consumption, obesity/ BMI. The investigators will also measure relevant variables of their clinical course such as regional block/anesthesia/epidural administration. Radiological appearance of presenting imaging (either CT Chest or chest X-ray) will be compared by a dedicated and blinded radiologist who will grade the initial imaging based on severity including the following variables: number of fractures, bilateral vs. unilateral, degree of displacement, presence of lung contusion, presence of pneumothorax, presence of intrinsic lung disease, pleural effusion or blood.

Survey results (both pretest and posttests) will be compared using the appropriate statistical methods depending on the questions construct: with Chi squared performed for categorical variables (such as multiple choice) and unpaired t test for continuous variables (such as likert scale rankings).

The investigators have performed a power calculation to determine if the following hypothesis can be reasonably answered with the trial of this size: the investigators hypothesize that the RibFx belt can improve pain control in the post-rib fracture setting for patients without impeding pulmonary functioning. The investigators anticipate seeing an improvement in pain scores and/or narcotic consumption within the rib belt group, without seeing significant differences in pulmonary function (although do expect a nonsignfiicant trend toward improved pulmonary function).

In order to perform our power function the investigators reviewed the literature to determine prior similar samples to our expected cohort. The investigators performed our power calculation with the goal of 80% power (with 2-sided alpha= 0.05). The investigators anticipate based on prior studies (Fabricant et al that the baseline chest wall pain score (MPQ PPI and MPQ PRI) were a median of 3 (range 0-5) and a mean of 28 +/- 16 (range 0-70) respectively1. Looking at a study for Bugaev et al, the investigators can also anticipate pain medicine requirements in the form of Mean Equianalgesic Dose (MED) of opioid pain medication. In this study, the MED for rib fracture patients was found to be 135.8 (IQR 50.83-440.0). Finally, Butts CA et al 3 studied incentive spirometry volume (ISV) scores in this population of patients and found their median ISV (in ml) was 1250 (IQR 750-1250).

For a one-group pre-post design, a sample size of 30 subjects would provide 83% power to detect a 20% decrease in MPQ PRI, assuming a within subject correlation of 0.8 for MPQ PRI scores and using a two-sided type I error rate of 0.05. A sample size of 35 (the planned size of the intervention group), provides an 88% power to detect a 20% decrease.

ELIGIBILITY:
Inclusion Criteria:

* Adult person age 18-80 admitted with at least one acute traumatic closed rib fracture to the University of Vermont Medical Center

Exclusion Criteria:

* Pediatric (<18 year old) and Geriatric (>80 year old) patients
* Patients who are intubated on arrival or within first 24 hours of admission or with Glasgow Coma Scale (GCS) < 14 (altered or depressed consciousness)
* Pregnant patients
* Patients who undergo operative rib fixation for their rib fractures (such as open reduction internal fixation, or rib plating)
* Patients with chest wall deformity, lacerations, burns, or soft tissue injuries that preclude placement of the RibFx belt
* Patients with an additional mechanism of injury that would create severe distracting pain, as determine by the admitting team.
* Isolated 1st rib or 2nd rib fractures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajai Malhotra, MD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: RibFx Belt Product Site — https://www.pelvicbinder.com/ribfx-belt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RibFx Belt Arm | Control
Started | 12 | 15
Completed | 11 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RibFx Belt Arm | Control | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 5 | 8 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 13 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Rib Fracture Subjective Self-Reported Pain (Inpatient)
Description: Compare pain control in patients with non-operatively managed traumatic rib fractures via subjective/qualitative self-reporting of pain control via questionnaires Pain control will be predominantly measured utilizing a likert scale score of 1 to 10, with a score of 1 denoting the lowest amount of pain and a score of 10 indicating the highest amount of pain. This will assist us in comparing patient pain scores in an objective manner.
Time Frame: Inpatient Stay
Population: Population described includes participants where data was collected regarding pain control during their inpatient stay (1 patient withdrawn prior to data collection).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RibFx Belt Arm | Control
Number analyzed (Participants) | 12 | 14
score on a scale | 5.96 (2.59) | 5.40 (1.85)

2. Primary Outcome: Narcotic/ Opioid Pain Medication Requirement After Rib Fracture (Inpatient)
Description: Count of participants who required any use of a prescribed pain medication at any point throughout their inpatient stay.
Time Frame: Inpatient Stay
Population: Population described includes participants where data was collected during inpatient stay (1 patient withdrawn prior to data collection).
Measure: Count of Participants; unit: Participants
Arm/Group | RibFx Belt Arm | Control
Number analyzed (Participants) | 12 | 14
Participants | 12 | 14

3. Secondary Outcome: Incentive Spirometry Score (Inpatient)
Description: Compare pulmonary hygiene and function amongst patients with non-operatively managed traumatic rib fractures via incentive spirometry scores.
  Incentive spirometry will be used as a tool to measure and compare patient pulmonary hygiene. The incentive spirometer at the participating institution are scaled to permit quantifiable deep breathing from 0 to 2500 mL (or cc).
Time Frame: Inpatient Stay
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | RibFx Belt Arm | Control
Number analyzed (Participants) | 12 | 14
mL | 1677.99 (688.55) | 1738.93 (575.38)

4. Secondary Outcome: Pneumonia Post Rib Fracture
Description: As measured by clinical diagnosis of pneumonia following rib fracture, either documented in physician note or added to problem list
Time Frame: 4 Week Follow Up
Population: Data not collected before study termination.
Arm/Group | RibFx Belt Arm | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Atelectasis Post Rib Fracture
Description: As measured by a participating blinded radiologist in any images obtained following the rib fractures
Time Frame: 4 Week Follow Up
Population: Data not collected before study termination.
Arm/Group | RibFx Belt Arm | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incentive Spirometry Score (Home)
Description: as for outcome 3
Time Frame: 4 Week Follow Up
Population: Population analyzed limited to those participants whose data was acquired through collection of home diary.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | RibFx Belt Arm | Control
Number analyzed (Participants) | 2 | 5
mL | 1693.75 (492.03) | 2028.75 (501.28)

7. Primary Outcome: Narcotic/ Opioid Pain Medication Requirement After Rib Fracture (Home)
Description: Count of participants who required any use of a prescribed pain medication at any point between their discharge from the hospital and their follow up appointment at 4 weeks.
Time Frame: 4 Week Follow Up
Population: Population analyzed limited to those participants whose data was acquired through administration of the questionnaire at their 4 week follow up appointment.
Measure: Count of Participants; unit: Participants
Arm/Group | RibFx Belt Arm | Control
Number analyzed (Participants) | 6 | 10
Participants | 3 | 3

8. Primary Outcome: Rib Fracture Subjective Self-Reported Pain (Home)
Description: as for outcome 1
Time Frame: 4 Week Follow Up
Population: Population analyzed limited to those participants whose data was acquired through completion of the follow up questionnaire at 4 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RibFx Belt Arm | Control
Number analyzed (Participants) | 6 | 10
score on a scale | 3.33 (2.80) | 3.30 (1.89)

ADVERSE EVENTS:
Time Frame: Date of Follow Up in Trauma Clinic (3-4 weeks)
Arm/Group | RibFx Belt Arm | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

LIMITATIONS AND CAVEATS:
This clinical trial was terminated on 5/25/2022 due to inadequate enrollment and data collection due to the COVID-19 pandemic. Of the 27 participants who were enrolled in the trial, only 5 patients yielded full data collection in all questionnaires/assessments. Other challenges including loss to follow up, discharge from the hospital before certain time points, and limited completion of the home log, all significantly limit our ability to analyze the data as intended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03846024/Prot_SAP_000.pdf